CLINICAL TRIAL: NCT01916382
Title: An International, Multicentre, Randomised, Evaluator-blind, No-treatment Controlled, Parallel-group Study to Assess the Efficacy and Safety of Once Daily Nitisinone in Patients With Alkaptonuria After 12 Months of Treatment, Followed by an Additional 36 Month Treatment Period.
Brief Title: Suitability of Nitisinone in Alkaptonuria 2
Acronym: SONIA 2
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Liverpool (Other)
Responsible Party: Principal Investigator, Professor Lakshminarayan Ranganath, Professor, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SONIA 2
Record Dates: First submitted 2013-08-02; First posted 2013-08-05 (Estimated); Last update posted 2018-05-31 (Actual); Status verified 2018-05

CONDITIONS: Alkaptonuria
Keywords: Alkaptonuria, nitisinone,Ochronosis, Homogentisic acid
MeSH Terms: conditions — Alkaptonuria; Ochronosis | interventions — nitisinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nitisinone (Experimental): Homogentisic acid lowering drug intervention
  Interventions: Drug: Nitisinone
- No treatment (No Intervention): comparrator

INTERVENTIONS:
Drug: Nitisinone — drug
  Other Names: Orfadin
  Arms: Nitisinone

SUMMARY:
This is a proposal to develop the orphan designated drug, nitisinone, for the treatment of a rare Mendelian disease, Alkaptonuria (AKU). Thanks to our existing successful fundamental and clinical research (cell models, animal models, natural history studies), we are now ready for this final stage of clinical development of nitisinone for AKU: a phase 3 clinical trial to prove efficacy. The results of DevelopAKUre will allow us to make the case to the European Medicines Agency for marketing authorisation of nitisinone for AKU, thereby contributing to the goal of the International Rare Diseases Research Consortium of developing 200 new therapies by 2020.

ELIGIBILITY:
Inclusion Criteria:

A patient must fulfil the following criteria in order to be included in the study:

1. Diagnosis of AKU Any Clinical manifestations of AKU, such as clinical ochronosis or chronic back/joint pain.

3. Age ≥25 years. 4. Willing and able to visit the investigational site for study visits. 5. Signed written informed consent given.

-

Exclusion Criteria:

The presence of any of the following will exclude a patient from inclusion in the study:

1. Currently pregnant or lactating.
2. Female patient of child-bearing potential not using a reliable method of contraception.
3. Known allergy to nitisinone or any of the constituents of the investigational product.
4. Current malignancy.
5. Uncontrolled hypertension (blood pressure greater than 180 mmHg systolic or greater than 95 mmHg diastolic).
6. Unstable cardiovascular disease.
7. Serum potassium < 3.0 mmol/L.
8. eGFR < 60 mL/min .
9. ALT > 1.5 x upper limit of normal.
10. Haemoglobin < 10.0 g/dL.
11. Platelets < 100 x 109/L.
12. Total white blood count < 3.0 x 109/L or neutrophil count < 1.5 x 109/L.
13. History of alcohol or drug abuse.
14. Participation in another clinical study within 3 months of randomization.
15. Treatment with nitisinone within 60 days of randomization.
16. Psychiatric or somatic illness that interferes with compliance or communication with health care personnel.
17. Foreseeable inability to cooperate with given instructions or study procedures.
18. Any other medical condition which in the opinion of the investigator makes the patient unsuitable for inclusion.

    -

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2020-02-02 (Estimated)

PRIMARY OUTCOMES:
24 houre Urine Homogentisic acid | year 1

CONTACTS AND LOCATIONS:
Overall Officials: L Ranganath, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Royal Liverpool Hospital, Liverpool, Merseyside, United Kingdom

REFERENCES:
- [Derived] Imrich R, Sedlakova J, Ulehlova M, Gornall M, Jackson R, Olsson B, Rudebeck M, Gallagher J, Lukacova O, Mlynarikova V, Stancik R, Vrtikova E, Zanova E, Zatkova A, Arnoux JB, Rovensky J, Luangrath E, Bygott H, Khedr M, Ranganath LR. Radiological evolution of spinal disease in alkaptonuria and the effect of nitisinone. RMD Open. 2022 Oct;8(2):e002422. doi: 10.1136/rmdopen-2022-002422. PMID 36270742
- [Derived] Ranganath LR, Psarelli EE, Arnoux JB, Braconi D, Briggs M, Broijersen A, Loftus N, Bygott H, Cox TF, Davison AS, Dillon JP, Fisher M, FitzGerald R, Genovese F, Glasova H, Hall AK, Hughes AT, Hughes JH, Imrich R, Jarvis JC, Khedr M, Laan D, Le Quan Sang KH, Luangrath E, Lukacova O, Milan AM, Mistry A, Mlynarikova V, Norman BP, Olsson B, Rhodes NP, Rovensky J, Rudebeck M, Santucci A, Shweihdi E, Scott C, Sedlakova J, Sireau N, Stancik R, Szamosi J, Taylor S, van Kan C, Vinjamuri S, Vrtikova E, Webb C, West E, Zanova E, Zatkova A, Gallagher JA. Efficacy and safety of once-daily nitisinone for patients with alkaptonuria (SONIA 2): an international, multicentre, open-label, randomised controlled trial. Lancet Diabetes Endocrinol. 2020 Sep;8(9):762-772. doi: 10.1016/S2213-8587(20)30228-X. Epub 2020 Aug 18. PMID 32822600